CLINICAL TRIAL: NCT01331772
Title: Randomized Controlled Study Assessing the Feasibility and the Medico-economic Impact of Nutritional Intervention in Women With Breast Cancer Under Adjuvant Chemotherapy
Brief Title: Impact of Nutritional Intervention in Women With Breast Cancer Under Adjuvant Chemotherapy
Acronym: PASAPAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Leon Berard (Other)
Collaborators: National Cancer Institute, France (Other Government); Ligue du Rhône (Unknown); Fondation de France (Other); Cancéropôle Lyon Auvergne Rhône-Alpes (Other); Lions Club Bourg-en-Bresse et Pérouges (Unknown); Association Lyonnaise de Logistique Posthospitalière (Other); Ministère de la Recherche (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: PASAPAS; 2011-A00064-37 (Other: AFSSAPS)
Record Dates: First submitted 2011-04-04; First posted 2011-04-08 (Estimated); Last update posted 2014-10-30 (Estimated); Status verified 2014-10

CONDITIONS: Breast Cancer; Adequate Physical Condition
Keywords: Breast cancer; Adapted Physical activity; Nutrition; Assessment; Patient education
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control arm (Other): Dietetic follow-up only
  Interventions: Other: Control arm
- Intervention arm (Experimental): Dietetic + adapted physical activity
  Interventions: Other: Intervention arm

INTERVENTIONS:
Other: Control arm — Dietetic follow-up only
  Arms: Control arm
Other: Intervention arm — Dietetic follow up + adapted physical activity
  Other Names: APA arm
  Arms: Intervention arm

SUMMARY:
Breast cancer is the most common cancer in women. Weight gain in adulthood, overweight or obesity, physical inactivity and alcohol consumption are risk factors commonly associated with risk of breast cancer (mainly for post-menopausal for overweight and obesity). Reduced physical activity is one factor likely to weight gain in women after adjuvant chemotherapy for localized breast cancer. Furthermore, physical activity appropriately could improve many prognostic factors and survival of women after breast cancer. Adapted Physical Activity (APA) could improve fitness, quality of life, body image, treatment compliance and reduce fatigue.

After diagnosis of breast cancer, there is many possible risk factors of mortality or morbidity related to nutritional factors available to management. These risks prevention through management of these patients appears indispensable through an APA program.

Thus, the investigators propose to test the feasibility of implementing a program of dietary intervention and APA to prevent the risk of weight gain (which affects more than half of patients) and maintain and/or increase their level of physical activity during and after adjuvant chemotherapy.

DETAILED DESCRIPTION:
With approximately 52,600 new cases diagnosed in France in 2010, breast cancer is the most common cancer in women, according to national projections of the incidence and cancer mortality for 2010.

Weight gain in adulthood, overweight or obesity, physical inactivity and alcohol consumption are risk factors commonly associated with risk of breast cancer (mainly for post-menopausal for overweight and obesity).

Several hypotheses explain the association between obesity and breast cancer: obesity, metabolic syndrome and diabetes participate to changes in hormone levels (estrogen, leptin, insulin) that promotes mammary carcinogenesis and tumor progression.

The association between obesity and development of breast cancer is partly due to increased serum levels of estradiol produced by adipocytes, but the role of insulin resistance and inflammation associated with obesity is widely discussed.

Reduced physical activity is one factor likely to weight gain in women after adjuvant chemotherapy for localized breast cancer. Furthermore, physical activity appropriately could improve many prognostic factors and survival of women after breast cancer. Thus, several large cohort studies of women with breast cancer showed an average mortality reduction of 45% associated with moderate physical activity compared with inactivity. Adapted Physical Activity (APA) could also improve fitness, quality of life, body image, treatment compliance and reduce fatigue.

A rich fruits and vegetables diet combined with regular physical activity appears to offer the best protection from breast cancer. The nature, frequency, duration, intensity and arrangement of physical training program meetings are key elements to consider, metabolic responses differ according to these factors.

The optimal management for an improved level of physical activity appear to be an individual of at least three sessions per week, 30 to 60 minutes each with a moderate intensity, allowing a physiological response to chronic exercise and an adequate recovery.

After diagnosis of breast cancer, there is thus many possible risk factors of mortality or morbidity related to nutritional factors available to management. These risks prevention through management of these patients appears indispensable through an APA program.

Thus, the investigators propose to test the feasibility of implementing a program of dietary intervention and APA to prevent the risk of weight gain (which affects more than half of patients) and maintain and/or increase their level of physical activity during and after adjuvant chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Female, 18 years ≤ age < 75 years
* With an invasive, non-metastatic, histologically confirmed, first breast carcinoma
* Requiring the prescription of a first line of adjuvant chemotherapy
* Followed in the research center
* Whose ability to participate in the APA intervention has been certified by a medical certificate issued by physician, the referring physician or the physician investigator
* Residing within a radius of 60 km around the center investigator or agreeing to bear the travel costs beyond proposed reimbursement
* Availability and willingness to invest in the PASAPAS study during the program (6 months) and during the post-program follow-up (6 months)
* Able to understand, read and write French
* Covered by a medical insurance
* Written, signed informed consent

Exclusion Criteria:

* Female with metastatic or inflammatory breast cancer,
* History or concomitant primary cancer (except for carcinoma in situ of the uterine cervix and/or skin basal cell carcinoma and or colon carcinoma in situ and/or not a breast cancer in complete response for at least 5 years)
* Cons-indication to physical activity practice, at discretion of the investigator,
* In a state of severe malnutrition according to the criteria of the High Authority for Health (HAS) 2010, namely:

  * Among women ≤ 70 years: weight loss ≥ 15% in 6 months or ≥ 10% in 1 month
  * Among women > 70 years: weight loss ≥ 15% in 6 months or ≥ 10% in 1 month, body mass index < 18 kg / m²
* History of eating disorders,
* Not possible follow-up for medical, social, familial, geographical or psychological reasons, during the program (6 months) and during the post-program follow-up (6 months),
* Deprived of their liberty by court or administrative decision,
* Pregnant or nursing, of childbearing age without effective contraception during the study.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2011-07; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Assessment in a cohort of adult patients with a 1st breast cancer non-metastatic, the feasibility of implementing an APA intervention during 6 months, in addition to a dietary management, concomitant to prescription of a first-line adjuvant chemotherapy | 6 months
  Proportion of patients who participate in at least two mandatory APA sessions by week during all the APA program, except during the 1st week of each course of CT

SECONDARY OUTCOMES:
Assessment of patients compliance to the implementation of the APA program and analyze of the reasons for noncompliance | 6 months
  Rate of patients who completed the full program and analysis of non-compliance grounds during the program
Assessment of acceptability of the intervention and randomization / recruiting capabilities | 6 months
  Number of patients contacted by the investigator to participate in the study and rate of patients randomized
Verification of adequacy between the conduct procedures of program (APA and dietetic) and the constraints of program implementing in real conditions | 12 months
  Formalization of a program used in real conditions
Description of patient satisfaction | Month 12
  Calculation of overall satisfaction score of patients on the treatment received, evaluated by a scale of satisfaction
Medico-economic impact of the intervention | 12 months
  Settlement expenses costs, incurred costs and costs avoided by the intervention
Biological study | Day 1 CT, week 9, week 24, month 12
  Analyses of metabolomic profiles and adipokines expression linked to breast cancer at initial diagnosis (before surgery) and description of metabolism changes during nutritional interventions and therapeutic care
Description of dietary | Day 1 CT, week 24, month 12
  Collection of patient nutritional intake during 3 days by self-administered questionnaire
Description of level and pattern physical activity | Day 1 CT, Week 9, Week 24, Month 12
  Evaluation of level and pattern physical evaluation (PAQAP and IPAQ questionnaire)
Description of anthropometry | Day 1 CT, week 9, week 24, month 12
  Measurement of weight, height, waist and hip circumference
Description of lipid profiles | Day 1 CT, week 9, week 24, month 12
  Measurement of total cholesterol, HDL, LDL and triglycerides
Assessment of life quality | Day 1 CT, week 24, month 12
  Life quality scores calculation (QLQ-C30, BR-23, MOS SF-36)
Description of anxiety | Day 1 CT, week 24, month 12
  score calculation of anxiety (STAI questionnaire)
Assessment of patients compliance to the implementation of diet and analyze of the reasons for noncompliance | 6 months
  Rate of patients who completed the full program and analysis of non-compliance grounds during the program
Description of body satisfaction | Day 1 CT, week 24, month 12
  score calculation of QSCPGS questionnaire
Description of body composition | Day 1 CT, week 9, week 24, month 12
  Measurement of body composition by impedancemetry
Description of self-perception | Day 1 CT, week 24, month 12
  score calculation of self-perception (QSCPGS questionnaire)
Description of self esteem | Day 1 CT, week 24, month 12
  score calculation of self-esteem (Rosenzweig scale)
Description of depression | Day 1 CT, week 24, month 12
  score calculation of depression (BDI questionnaire)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick BACHMANN, MD, Principal Investigator — Centre Leon Berard
Locations (1):
- Centre Leon Berard, Lyon, France

REFERENCES:
- [Result] Majed B, Moreau T, Senouci K, Salmon RJ, Fourquet A, Asselain B. Is obesity an independent prognosis factor in woman breast cancer? Breast Cancer Res Treat. 2008 Sep;111(2):329-42. doi: 10.1007/s10549-007-9785-3. Epub 2007 Oct 16. PMID 17939036
- [Result] Tredan O, Bajard A, Meunier A, Roux P, Fiorletta I, Gargi T, Bachelot T, Guastalla JP, Lallemand Y, Faure C, Perol D, Bachmann P. Body weight change in women receiving adjuvant chemotherapy for breast cancer: a French prospective study. Clin Nutr. 2010 Apr;29(2):187-91. doi: 10.1016/j.clnu.2009.08.003. Epub 2009 Aug 26. PMID 19713014
- [Result] Holmes MD, Chen WY, Feskanich D, Kroenke CH, Colditz GA. Physical activity and survival after breast cancer diagnosis. JAMA. 2005 May 25;293(20):2479-86. doi: 10.1001/jama.293.20.2479. PMID 15914748
- [Result] Newton RU, Galvao DA. Exercise in prevention and management of cancer. Curr Treat Options Oncol. 2008 Jun;9(2-3):135-46. doi: 10.1007/s11864-008-0065-1. Epub 2008 Aug 13. PMID 18704691
- [Result] Pierce JP, Stefanick ML, Flatt SW, Natarajan L, Sternfeld B, Madlensky L, Al-Delaimy WK, Thomson CA, Kealey S, Hajek R, Parker BA, Newman VA, Caan B, Rock CL. Greater survival after breast cancer in physically active women with high vegetable-fruit intake regardless of obesity. J Clin Oncol. 2007 Jun 10;25(17):2345-51. doi: 10.1200/JCO.2006.08.6819. PMID 17557947
- [Derived] Febvey-Combes O, Jobard E, Rossary A, Pialoux V, Foucaut AM, Morelle M, Delrieu L, Martin A, Caldefie-Chezet F, Touillaud M, Berthouze SE, Boumaza H, Elena-Herrmann B, Bachmann P, Tredan O, Vasson MP, Fervers B. Effects of an Exercise and Nutritional Intervention on Circulating Biomarkers and Metabolomic Profiling During Adjuvant Treatment for Localized Breast Cancer: Results From the PASAPAS Feasibility Randomized Controlled Trial. Integr Cancer Ther. 2021 Jan-Dec;20:1534735420977666. doi: 10.1177/1534735420977666. PMID 33655799
- [Derived] Perrier L, Foucaut AM, Morelle M, Touillaud M, Kempf-Lepine AS, Heinz D, Gomez F, Meyrand R, Baudinet C, Berthouze S, Reynes E, Carretier J, Guillemaut S, Perol D, Tredan O, Philip T, Bachmann P, Fervers B. Cost-effectiveness of an exercise and nutritional intervention versus usual nutritional care during adjuvant treatment for localized breast cancer: the PASAPAS randomized controlled trial. Support Care Cancer. 2020 Jun;28(6):2829-2842. doi: 10.1007/s00520-019-05078-4. Epub 2019 Nov 15. PMID 31729566
- [Derived] Foucaut AM, Morelle M, Kempf-Lepine AS, Baudinet C, Meyrand R, Guillemaut S, Metzger S, Bourne-Branchu V, Grinand E, Chabaud S, Perol D, Carretier J, Berthouze SE, Reynes E, Perrier L, Rebattu P, Heudel PE, Bachelot T, Bachmann P, Fervers B, Tredan O, Touillaud M. Feasibility of an exercise and nutritional intervention for weight management during adjuvant treatment for localized breast cancer: the PASAPAS randomized controlled trial. Support Care Cancer. 2019 Sep;27(9):3449-3461. doi: 10.1007/s00520-019-4658-y. Epub 2019 Jan 24. PMID 30680617